CLINICAL TRIAL: NCT05875038
Title: Superiority of Intelligent Video Surveillance + Telealarm Over Telealarm Alone in Elderly People at Risk of Falling
Acronym: VIGIALARM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Hôpital Les Bateliers, CHU de Lille (Unknown); Hôpital cardiologique, CHU de Lille (Unknown); Hôpital Saint Philibert, GHICL (Unknown); Hôpital Côte de Nacre, CHU de Caen (Unknown); Hopital Charles Nicolle (Other); University Hospital, Rouen (Other); Centre Hospitalier de Saint-Quentin (Unknown); Centre Hospitalier de Beauvais (Other); Centre Hospitalier de Valenciennes (Network); CHU Peronne (Unknown); Centre Hospitalier de l'Arrondissement de Montreuil-sur-mer (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI2019_843_0062
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Intelligent Video Surveillance; Fall; Home; Frail Elderly Person
Keywords: intelligent video surveillance; Fall; home; frail elderly person; teleassistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intelligent Video Monitoring + Tele-alarm (Experimental)
  Interventions: Other: video system; Other: Tele-alarm
- Tele-alarm only (Active Comparator)
  Interventions: Other: Tele-alarm

INTERVENTIONS:
Other: video system — The video surveillance system will analyze the position of subjects in real time using algorithms based on artificial intelligence. The system works continuously without video capture and sends an alert with a photo if a person is lying down after a fall. The alert is confirmed after an operator has checked the photo capture on a dedicated platform.
  Arms: Intelligent Video Monitoring + Tele-alarm
Other: Tele-alarm — Tele-alarm

SUMMARY:
Maintaining the elderly at home and preventing them from falling are major public health issues. The vast majority of elderly people wish to remain at home. The fear of a fall with prolonged standing is a frequent reason for institutionalization. There are few procedures that have been shown to be effective in preventing falls and their complications. Prolonged standing on the floor is a major complication that can lead to multiple events, including death.

Tele-alarms are widely used in France and in Europe, but their effectiveness in the event of a fall is poor and their use is restrictive (they require physical and mental capacities to activate). However, elderly people at risk of falling are often frail or dependent, suffering from cognitive disorders and sometimes polymorbid, which explains the large number of failures of tele-alarms. There are other alert systems, notably intelligent video surveillance systems such as the VA2CS. This is a video system placed in the home that analyzes the position of subjects in real time using algorithms based on artificial intelligence. The system works continuously without video capture and sends an alert with a photo if a person is lying down after a fall. The alert is confirmed after an operator has checked the photo capture on a dedicated platform. To date, it has a sensitivity and specificity of over 90% (manufacturer's data not published). Its performance is equivalent to other intelligent video surveillance systems published in the literature. This system is autonomous and does not rely on the abilities of the person at risk of falling. Intelligent video surveillance is an innovative technology which has not yet been evaluated in a geriatric care program, nor compared to a reference or analyzed from a quality of life or medico-economic perspective.

The hypothesis of this study is that intelligent video surveillance allows an exhaustive and early detection of the fall with a faster alert enabling to avoid prolonged standing on the ground and its consequences compared to the tele-alarm alone.

ELIGIBILITY:
Inclusion Criteria:

* Person aged 75 years or more
* hospitalized in an acute geriatric service or in a geriatric or multipurpose rehabilitation care service
* If living alone: receiving at least one visit per day from a relative or professional
* Recent history of fall and monopodal support < 5 seconds
* Able to give informed consent.
* Return home considered complex by the patient or their relatives due to the risk of falling at home.

Exclusion Criteria:

* Under legal protection
* Not affiliated to a social security system
* Confined to bed or chair

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 395 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of at least one unscheduled rehospitalization | 90 days
  Occurrence of at least one unscheduled rehospitalization within the first 90 days following the return home.

SECONDARY OUTCOMES:
number of days during unscheduled hospitalization | 90 days
  number of days during unscheduled hospitalization
Number of days in emergency | 90 days
  Number of days in emergency within the first 90 days following the return home

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No